CLINICAL TRIAL: NCT00080678
Title: Randomized Double-Blind Phase II Trial of Docetaxel and Imatinib Versus Docetaxel and Placebo in Metastatic Androgen-Independent Prostate Cancer (AIPC) With Bone Metastases
Brief Title: Docetaxel With or Without Imatinib Mesylate in Treating Patients With Androgen-Independent Prostate Cancer and Bone Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000354505; MDA-ID-030008; NOVARTIS-MDA-ID-030008; MSKCC-03132; DFCI-03187
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Docetaxel; Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel + Imatinib Mesylate (Experimental): Docetaxel 30 mg/m^2 intravenous over 60 minutes on days 1, 8, 15, and 22 in 42-day cycles, with daily oral 600 mg imatinib mesylate.
  Interventions: Drug: Docetaxel; Drug: Imatinib Mesylate
- Docetaxel + Placebo (Placebo Comparator): Docetaxel 30 mg/m^2 intravenous (IV) over 60 minutes on days 1, 8, 15, and 22 in 42-day cycles, with daily oral placebo.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel
  Other Names: taxotere
Drug: Imatinib Mesylate
  Other Names: Imatinib; Gleevec; STI571; NSC-716051
  Arms: Docetaxel + Imatinib Mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining docetaxel with imatinib mesylate may be effective treatment for androgen-independent prostate cancer and bone metastases.

PURPOSE: This randomized phase II trial is studying docetaxel and imatinib mesylate to see how well they work compared to docetaxel alone in treating patients with androgen-independent prostate cancer and bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to progression in patients with androgen-independent prostate cancer and bone metastases treated with docetaxel with vs without imatinib mesylate.

Secondary

* Compare the response rates in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to hemoglobin (< 11g/dL vs ≥ 11 g/dL), alkaline phosphatase (normal vs elevated), number of prior regimens (0 vs 1 or 2), and ECOG performance score (0 or 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV on days 1, 8, 15, and 22 and oral imatinib mesylate once daily on days 1-43.
* Arm II: Patients receive docetaxel as in arm I and oral placebo once daily on days 1-43.

In both arms, courses repeat every 43 days in the absence of disease progression or unacceptable toxicity. Patients who progress on arm II may cross over to arm I.

PROJECTED ACCRUAL: A total of 152 patients (76 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate

  * Osseous metastases confirmed by radiography
  * Lytic bone lesions considered for biopsy if there is clinical suspicion of histologic conversion to small cell carcinoma
* Failed prior hormonal therapy
* Progressive disease, as evidenced by one of the following:

  * 2 consecutive rises in prostate-specific antigen (PSA) of at least 1 ng/mL over 4 weeks
  * Increase of 25% of the product of bidimensional disease or 30% in maximum diameter
  * Increase in number of osseous metastases by bone scan
  * Worsening symptoms attributable to disease progression (e.g., worsening bony pain)
* PSA ≥ 1 ng/mL
* Castrate serum testosterone ≤ 50 ng/dL

  * Concurrent luteinizing-hormone releasing-hormone analog required for medically castrated patients
* No small cell or sarcomatoid prostate cancers
* No uncontrolled CNS metastases

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤ 2 times upper limit of normal
* No chronic liver disease

Renal

* Creatinine clearance ≥ 40 mL/min

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No unstable angina
* No myocardial infarction within the past 6 months
* No evidence of myocardial ischemia on electrocardiogram
* No uncontrolled severe hypertension

Pulmonary

* No oxygen-dependent lung disease

Other

* HIV negative
* No concurrent severe infection
* No contraindication to corticosteroids
* No uncontrolled diabetes mellitus
* No grade 2 or greater peripheral neuropathy
* No other malignancy within the past 2 years except nonmelanoma skin cancer
* No overt psychosis, mental disability, or incompetency that would preclude giving informed consent
* No history of noncompliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior taxanes
* No more than 2 prior chemotherapy regimens
* At least 30 days since prior chemotherapy and recovered
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior flutamide or nilutamide*
* At least 6 weeks since prior bicalutamide* NOTE: *Unless there is evidence of interim disease progression

Radiotherapy

* At least 90 days since prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium and recovered
* At least 30 days since other prior radiotherapy and recovered

Surgery

* Fully recovered from prior surgery

Other

* No concurrent ketoconazole
* No concurrent warfarin

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2003-05; Primary Completion 2005-08 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Time to progression | Baseline to 3 years, or until disease progression

SECONDARY OUTCOMES:
Response rate | Up to 3 years
Toxic effects | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, Study Chair — M.D. Anderson Cancer Center; Christopher Logothetis, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Result] Mathew P, Thall PF, Johnson MM, et al.: Preliminary results of a randomized placebo-controlled double-blind trial of weekly docetaxel combined with imatinib in men with metastatic androgen-independent prostate cancer (AIPC) and bone metastases (BM). [Abstract] J Clin Oncol 24 (Suppl 18): A-4562, 232s, 2006.